CLINICAL TRIAL: NCT01335295
Title: Open Pilot Trial to Test the Safety and Tolerability of Flavocoxid in Duchenne Muscular Dystrophy
Brief Title: Safety Study of Flavocoxid in Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Giuseppe Vita, full professor, University of Messina
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DMD-2011
Record Dates: First submitted 2011-04-12; First posted 2011-04-14 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Flavocoxid; Duchenne muscular dystrophy; pilot study
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — flavocoxid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Flavocoxid — Flavocoxid capsules TTD 500 mg/die or 1000 mg/die for 1 year

SUMMARY:
Objective of this study is to evaluate safety and tolerability of flavocoxid administered at the daily oral dose of 500 or 1000 mg/die for one year in DMD patients, alone or in association with steroids (deflazacort on alternate days) started at least one year before. The investigators will also perform a multidimensional clinical evaluation covering functional and muscle strength and quality of life (QoL)assessments.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of DMD, confirmed by muscle biopsy and molecular analysis by MPLA;
* range of age between 4 -16 years;
* unaided ambulation for at least 75 meters, unassisted during the Screening 6MWT. Other personal assistance or use of assistive devices for ambulation (eg, short leg braces, long leg braces or walkers) is not permitted.
* follow-up of at least 1 year before baseline with the selected motor outcome measures;
* patients able to perform evaluation tests;
* patient legally authorized representative (LAR) able to understand and give the informed consent;
* absence of contra-indications to the use of flavocoxid (see below);
* written informed consent signed by LAR.

Exclusion Criteria:

* treatment with other drugs analogue, similar or interacting with flavocoxid or immunosuppressive therapy (other than corticosteroids) within 3 months prior to start of study treatment;
* exposure to another investigational drug or supplements within 2 months prior to start of study treatment;
* presence of cognitive impairment that could influence the performance of the evaluation tests;
* history of major surgical procedure within 30 days prior to start of study treatment;
* expectation of major surgical procedure (eg, scoliosis surgery) during the 12-month treatment period of the study;
* ongoing participation in any other therapeutic clinical study;
* expectation of recruitment in the forthcoming exon-51 trial;
* requirement for daytime ventilator assistance;
* presence of liver-diseases or assumption of any hepatotoxic agent;
* screening laboratory values out of the laboratory ranges if clinically meaningful;
* prior or ongoing medical condition (eg, concomitant illness, psychiatric condition, behavioral disorder, alcoholism, drug abuse), medical history, physical findings, ECG findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the subject, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.

Ages: 4 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
All adverse events and laboratory or ECG abnormalities | 1 year

SECONDARY OUTCOMES:
Motor assessments and biochemical evaluation | 1 year
  Outcome measures will include:
  * Functional tests: 6- minute walk test, North Star Ambulatory Assessment (NSAA) with timed items
  * Medical Research Council (MRC) score of upper and lower limbs;
  * Maximum voluntary isometric contraction (MVIC)
  * Quality of Life (QoL) evaluation ;
  * Forced vital capacity (FVC) with spirometer . Changes in biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Vita, MD, Principal Investigator — Department of Neuroscience, University of Messina
Locations (1):
- Department of Neuroscience, Psychiatry and Anestesiology, Policlinico of Messina, Messina, ME, Italy